CLINICAL TRIAL: NCT02176070
Title: Reproductive Health in Men and Women With Vasculitis
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Duke University (Other); Boston University (Other); Data Management and Coordinating Center (DMCC) (Other)
Responsible Party: Sponsor
Other Study IDs: 5531
Record Dates: First submitted 2014-05-30; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Giant Cell Arteritis; Takayasu's Arteritis; Polyarteritis Nodosa; Wegener's Granulomatosis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Behcet's Disease; Kawasaki Disease; Henoch-schoenlein Purpura; Vasculitis, Central Nervous System; Drug-induced Necrotizing Vasculitis
MeSH Terms: conditions — Giant Cell Arteritis; Takayasu Arteritis; Polyarteritis Nodosa; Granulomatosis with Polyangiitis; Microscopic Polyangiitis; Churg-Strauss Syndrome; Behcet Syndrome; Mucocutaneous Lymph Node Syndrome; IgA Vasculitis; Vasculitis, Central Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to learn about reproductive health, including fertility and pregnancies, in people with vasculitis.

DETAILED DESCRIPTION:
All patients enrolled in the Vasculitis Clinical Research Consortium's Contact Registry were invited via email to participate in this study. The Contract Registry includes people who self-identify as having one of 6 vasculitities: Wegener's Granulomatosis, Microscopic Polyangiitis, Churg-Strauss Syndrome, Polyarteritis Nodosum, Takayasu's Arteritis, and Giant Cell Arteritis. People voluntarily enroll in this Registry with the understanding that they will receive information about clinical studies for which they might be eligible. The introductory email included basic information about the study and all of the required elements for informed consent in a brief format. By clicking the link to the reproductive health questionnaire, participants gave their consent to be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in VCRC Contact Registry
* Patient reported diagnosis of Wegener's Granulomatosis, Microscopic Polyangiitis, Churg-Strauss Syndrome, Polyarteritis Nodosa, Takayasu's Arteritis, Giant Cell Arteritis, Behcet's Disease, Kawasaki Disease, Henoch-Schoenlein Purpura, CNS or Drug-induced Vasculitis
* 18 years of age or older
* English speaking

Exclusion Criteria:

* Inability to provide informed consent and complete survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with vasculitis included in the VCRC Contact Registry were invited to participate. Data was included for all patients who provided a vasculitis diagnosis, estimated date of diagnosis, confirmed that the diagnosis was made by a rheumatologist, and reported having taken at least one appropriate anti-rheumatic medication. Other participants were excluded as the likelihood that they have a true vasculitis condition is low.
Sampling Method: Non-Probability Sample
Enrollment: 467 (Actual)
Dates: Start 2011-02; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The rate of infertility with and without prior cyc. | 1 year after the study is closed to enrollment

SECONDARY OUTCOMES:
The rate of pregnancy complications in pregnancies delivered before and after vasculitis diagnosis. | 1 year after the study is closed to enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Megan Clowse, MD, MPH, Study Chair — Duke University; Amanda M. Terry, MA, Study Chair — USF College of Medicine
Locations (1):
- University of South Florida Data Management Coordinating Center, Tampa, Florida, United States